CLINICAL TRIAL: NCT03701347
Title: A Comparison of Three Simulators for Colposcopy LEEP Training
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, Ida Suzani Ismail, Instructor, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: S-18-072E
Record Dates: First submitted 2018-09-30; First posted 2018-10-10 (Actual); Last update posted 2018-10-12 (Actual); Status verified 2018-09

CONDITIONS: Colposcopy
Keywords: Colposcopy; Simulator; Comparison Study; Learning effectiveness

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Reeve's model (Active Comparator): After introduction of Loop excision electrosurgical procedure through video, participants will undergo Reeve's simulators
  Interventions: Device: Reeve's model
- Hefler's model (Active Comparator): After introduction of Loop excision electrosurgical procedure through video, participants will undergo Hefler's simulators
  Interventions: Device: Hefler's model
- Ida's Model (Experimental): After introduction of Loop excision electrosurgical procedure through video, participants will undergo Ida's simulators
  Interventions: Device: Ida's model

INTERVENTIONS:
Device: Reeve's model — Reeves, K. O., Young, A. E., & Kaufman, R. H. (1999). A simple, inexpensive device for teaching the loop electrosurgical excision procedure. Obstetrics and Gynecology, 94(3), 474-5.
  Arms: Reeve's model
Device: Hefler's model — Hefler, L., Grimm, C., Kueronya, V., Tempfer, C., Reinthaller, A., & Polterauer, S. (2012). A novel training model for the loop electrosurgical excision procedure: An innovative replica helped workshop participants improve their LEEP. American Journal of Obstetrics and Gynecology, 206(6)
  Arms: Hefler's model
Device: Ida's model — Reusable, portable and modular 3D printed simulator
  Arms: Ida's Model

SUMMARY:
This randomized controlled trial evaluates the learning effectiveness of three different types of Colposcopy simulators objectively with Objective Structured Assessment of Technical Skill (OSATS) and subjectively with self-reported confidence survey. A total of 60 participants, randomly assigned into 3 groups, will learn from Hefler's, Reeve's or authors' simulators. The investigators hypothesize that the proposed simulator affords better learning objectively and subjectively with improved functional fidelity.

DETAILED DESCRIPTION:
Colposcopy and colposcopic treatment is a unique skill that is acquired only following careful training. A colposcopist plays an important role to correctly diagnose, take appropriate biopsies and perform appropriate safe and effective treatment of women with preinvasive cervical disease. However, no surgical treatment comes without risk and colposcopy treatment is no different. Risks from a colposcopy treatment can include intraoperative complication such as bleeding, injury to surrounding organs by the instrument used i.e. laser burns, diathermy burns and damage to bladder, rectum, vulva or vagina. Other complication may include insufficient tissue excised or ablated during treatment leading to failure of cure and risk of recurrent treatment. Recurrent treatment especially excisional treatment has been shown to increase the risk of preterm labour for future pregnancies. In view of this, training in colposcopy and colposcopy treatment is a crucial part of effective cervical cancer prevention.

In this study, the investigators aim to determine if Hefler's, Reeve's or authors' simulators are more effective at supporting the colposcopy training. The significance of the result lies in the effectiveness of training simulator for colposcopy training and the confidence of doctors when they perform their first colposcopy.

ELIGIBILITY:
Inclusion Criteria:

* Year 4 and Year 5 Medical students who have completed their Obstetrics and gynaecology attachment
* Practicing medical doctors who have and have not performed Colposcopy LEEP

Exclusion Criteria:

* Students who have not completed their Obstetrics and gynaecology attachment

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-09-29 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
OSATS Score | 10 minutes
  Objective structured assessment of technical skills (OSATS) scores rose before and after completion of training
  Competency Scale. Score of 2 indicates participant can performed task independently.Score of 1 indicates participant need help performing task. Score of 0 indicates participant has not performed the task.
  1. Use of speculum
  2. Using Colposcope for good visualization of area to be excised.
  3. Infiltration of local anaesthetic: adrenaline circumferentially around lesion to be
  4. excised using the dental syringe provided.
  5. Perform LEEP in 1 single pass producing 1 specimen only.
Self-reported confidence score | 1 minute
  Likert scale of 1 to 5. Score of 1 indicates very low confidence whereas a score of 5 indicates high confidence at performing the procedures.

SECONDARY OUTCOMES:
Quality of specimen | 10 minutes
  Blinded assessor using validated scoring system. Score of 1 indicates very poor techniques whereas a score of 5 indicates clearly superior techniques.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics & Gyanecology, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No